CLINICAL TRIAL: NCT01190631
Title: An Assessment of Residual Spherical Aberration, Postoperative Total High Order Aberrations, and Functional Vision Correlation After SN60WF IOL Implantation
Brief Title: An Assessment of Residual Spherical Aberration, Postoperative Total High Order Aberrations, and Functional Vision Correlation Following Intraocular Lens (IOL) Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M-10-008
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Cataracts
Keywords: intraocular lens; cataracts; total residual spherical aberration; high order aberrations
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acrysof IQ (SN60WF) IOL (Experimental): AcrySof IQ SN60WF intraocular lens (IOL) implanted in one eye only during cataract surgery.
  Interventions: Device: Acrysof IQ (SN60WF) IOL

INTERVENTIONS:
Device: Acrysof IQ (SN60WF) IOL — Acrysof IQ (SN60WF) intraocular lens implanted in the capsular bag of the eye during cataract surgery. The IOL is intended for the lifetime of the patient. Unilateral (one eye only) implantation is planned.
  Other Names: Acrysof® IQ Model SN60WF

SUMMARY:
The purpose of this study was to evaluate total residual spherical aberration (TSA) post-IOL implantation, and to determine if an association exists between TSA, postoperative high order aberrations (HOA), and functional vision following IOL implantation in patients grouped by pre-operative corneal spherical aberration (CSA).

DETAILED DESCRIPTION:
Patients will be grouped by pre-operative corneal spherical aberration (CSA) measures, i.e., ≤0.230 micron and ≥0.270 micron.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract grade 3 or lower in at least one eye;
* Planned cataract removal via phacoemulsification with an implantation of an aspheric IOL;
* Able to have an operation within 30 days of preoperative evaluation;
* Good ocular health, with the exception of cataracts;
* ≤ 1.50 diopter (D) of preoperative astigmatism by keratometry;
* Willing and able to understand and sign an informed consent;
* Willing and able to attend postoperative examinations per protocol schedule;
* Able to achieve 6.5mm dilated pupil;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Preoperative ocular pathology as specified in protocol;
* Preoperative corneal pathology as specified in protocol;
* Keratometric astigmatism exceeding 1.50 diopter;
* Planned postoperative refraction for mono-vision;
* Uncontrolled diabetes;
* Use of any systemic or topical drug known to interfere with visual performance;
* Contact lens use during the active treatment portion of the trial;
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis;
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results;
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial;
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye;
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control;
* Other protocol-defined exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Contrast Sensitivity | Day 90 postoperative
  Contrast sensitivity is the measurement of one's ability to detect slight changes in luminance before it becomes indistinguishable. It is measured in logarithmic units by means of an illuminated box, the CSV 1000 by Vector Vision. A higher value for the logarithmic units translates to better contrast sensitivity.

SECONDARY OUTCOMES:
Total Higher Order Aberrations | Day 90 postoperative
  A higher order aberration is a distortion acquired by a wavefront light when it passes through an eye with irregularities of its refractive components (tear film, cornea, aqueous humor, crystalline lens and vitreous humor). It is measured via wavefront measurements according to manufacturer's instructions with a LADARWave (Alcon Laboratories, Inc., Ft. Worth TX).
Corneal Spherical Aberration | Day 90 postoperative
  Corneal spherical aberration is the blurring of an image that occurs when light from the margin of a lens or mirror with a spherical surface comes to a shorter focus than light from the central portion. The changing focal length is caused by deviations in the lens or mirror surface from a true sphere and is measured by corneal topography with a commercially available topographer in accordance with manufacturer's guidelines.
Uncorrected Visual Acuity (UCVA) | Day 90 postoperative
  Uncorrected visual acuity, i.e., visual acuity without any type of corrective lenses, is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution," and a lower logMAR value indicates better visual acuity.
Best Corrected Visual Acuity (BCVA) | Day 90 postoperative
  Best corrected visual acuity, i.e., visual correction utilizing a phoropter or trial frames, is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution," and a lower logMAR value indicates better visual acuity.
Low Contrast (10%) Visual Acuity | Day 90 postoperative
  Visual acuity is tested using 10% contrast ETDRS (Early Treatment Diabetic Retinopathy Study) charts under photopic conditions. Testing is performed using the correction from the manifest refraction at a distance calibrated for the chart. Visual acuity (VA) is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution," and a lower logMAR value indicates better visual acuity.
Quality of Vision Questionnaire | Day 90 postoperative
  As completed by the participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States